CLINICAL TRIAL: NCT05239754
Title: Fresno Area Workforce Development Board Family-Focused, Interconnected, Resilient, Essential Healthy Marriage and Responsible Fatherhood Program Evaluation
Brief Title: Fresno FAWDB FIRE Program Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Evaluation & Research (Other)
Collaborators: Fresno Area Workforce Development Board (FAWDB) (Unknown)
Responsible Party: Principal Investigator, Matt Shepherd, Principal Investigator, Midwest Evaluation & Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2021/03/39
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Results first posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Fathers

STUDY DESIGN:
Intervention Model Description: Arms Primary services: Participants receive 16 hours of 24/7 Dads curricula and at least 2 hours of career readiness workshops over the course of 9 weeks. Participants also receive ongoing job readiness support and post-employment support.
  Assigned Interventions Primary services: Participants receive 16 hours of 24/7 Dads curricula and at least 2 hours of career readiness workshops over the course of 9 weeks. Participants also receive ongoing job readiness support and post-employment support.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Primary Services (Experimental): Primary services: Participants receive 16 hours of 24/7 Dads curricula and at least 2 hours of career readiness workshops over the course of 9 weeks. Participants also receive ongoing job readiness support and post-employment support.
  Interventions: Other: Primary Services

INTERVENTIONS:
Other: Primary Services — Primary services: Participants receive 16 hours of 24/7 Dads curricula and at least 2 hours of career readiness workshops over the course of 9 weeks. Participants also receive ongoing job readiness support and post-employment support.

SUMMARY:
The purpose of the Fresno Area Workforce Development Board FIRE program evaluation is to determine whether primary (i.e., behaviors) and secondary (i.e., attitudes) outcomes improve for participants after completing the Fresno FIRE program. Understanding the ways in which the Fresno FIRE program supports healthy parenting relationships and financial stability is important for those providing services to at-risk fathers.

DETAILED DESCRIPTION:
After being informed about the study and giving consent, participants will enroll in a nine-week Fresno Fatherhood program that collects data at enrollment, at the end of the program, and 12 months following the program. Research questions in this study are framed by a descriptive evaluation design to assess whether outcomes improve for low-income fathers who participate in the Fresno FIRE program. Primary and secondary outcomes are assessed before and after participants complete core curricula - 24/7 Dads and career readiness workshops (pre to post). Primary outcome measures will indicate whether behavior improved for healthy family relationships (parent, co-parent, and partner) and economic stability (financial, employment). Secondary outcomes will indicate whether improvements were made in the attitudes and expectations that facilitate and reflect behavior for healthy family relationships and economic stability.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age 18 and older)
* Father/father figure of child under 24 years of age
* Residing in Fresno area, CA
* Has at-risk factors (residing in high poverty area, formerly justice-involved)

Exclusion Criteria:

* Minor (under the age of 18)
* Not a father/father figure
* Father of a child over 24 years of age
* Reside outside of Fresno area, CA

Min Age: 18 Months | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Father or father-figure
Enrollment: 488 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt D Shepherd, PhD, Principal Investigator — Midwest Evaluation & Research
Locations (1):
- Fresno Areas Workforce Development Board, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be confidential and aggregated. No individual participant data will be released unless requested by the courts. This study looks at data as a whole.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Services
Started | 488
Completed | 488
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Primary Services
Number analyzed (Participants) | 488
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 485
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 37.26 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 488
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 49
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 10
  Black or African American | 88
  White | 137
  More than one race | 186
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Healthy Parenting Behavior Measurement #1
Description: 1A) Will Fresno Fatherhood program participants experience significant increases in healthy parenting behaviors one year after program enrollment?
  Items measured include:
  Parenting behavior and interaction with children measured with:
  9 items- frequency of engagement in key behaviors (categories, 5-point scale)
  Measured on the Healthy Parenting Behavior Scale #1 as:
  1=Never 2=1 to 2 days per month 3=3 or 4 days per month 4=2 or 3 days per week 5=Every day or almost every day
  Higher ratings indicate higher frequency of engagement in parenting behavior and interaction with children, so the higher the rating, the better the score.
  The 9 items are measured as a construct. All items are added together and divided by 9 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: Change from baseline in behavior in parenting behavior (interaction with children at 12 months from enrollment).]
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 104
score on scale
  mean at baseline | 3.67 (1.022)
  mean at follow-up | 4.10 (0.830)

2. Primary Outcome: Healthy Co-parenting Behavior Measurement #1
Description: Will Fresno Fatherhood program participants experience significant increases in healthy co-parenting behaviors one year after program enrollment?
  Items measured include:
  Co-parenting behavior measured with:
  11 items: frequency of agreement with key co-parenting behaviors (interval, 5-point scale)
  Measured on the Healthy Co-Parenting Behavior Scale #1 as:
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  The 11 items are measured as a construct. All items are added together and divided by 11 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: Change from baseline in co-parenting behavior at 12 months from enrollment.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 267
score on scale
  mean at baseline | 3.49 (1.04)
  mean at follow-up | 3.50 (1.01)

3. Primary Outcome: Healthy Financial Behavior Measurement #1
Description: Will Fresno Fatherhood program participants experience significant increases in healthy financial behaviors one year after program enrollment?
  Items measured include:
  Father financial behavior measured with:
  2 items: yes (1) or no (0) questions for have checking account and have a savings account (dichotomous)
  Yes (1) responses indicate financial readiness, so the higher the rating, the better the score.
Time Frame: Change in parenting attitudes (towards children) at 12 months from enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Services
Number analyzed (Participants) | 329
Participants
  have savings account-baseline | 71
  have savings account-follow-up | 105
  have checking account-baseline | 76
  have checking account-follow-up | 137

4. Secondary Outcome: Healthy Parenting Attitudes Measurement #1
Description: Will Fresno Fatherhood program participants experience significant increases in healthy parenting attitudes/beliefs/expectations after completing the Fresno Fatherhood program?
  Items measured include:
  Parenting attitudes toward children measured with:
  7 items: frequency of key attitudes (categories, 5-point scale)
  Measured on the Healthy Parenting Attitudes Scale #1 as:
  1. Always
  2. Often
  3. Sometimes
  4. Rarely
  5. Never
  The 7 items are measured as a construct. All items are added together and divided by 7 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0.
Time Frame: Change in parenting attitudes (towards children) from baseline to immediately after program completion.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 225
score on scale
  mean at baseline | 4.55 (.482)
  mean at follow-up | 4.57 (.451)

5. Secondary Outcome: Healthy Financial Attitudes
Description: Will Fresno Fatherhood program participants experience significant increases in healthy financial attitudes/beliefs/expectations after completing the Fresno Fatherhood program?
  Items measured include:
  7 items: agreement with key financial attitudes (categories, 5-point scale)
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  The 7 items are measured as a construct. All items are added together and divided by 7 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: Change in healthy financial attitudes from baseline to immediately after program completion.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 418
score on scale
  mean at baseline | 3.46 (.603)
  mean at follow-up | 3.64 (.635)

6. Secondary Outcome: Healthy Employment Behaviors
Description: Will Fresno Fatherhood program participants experience significant increases in healthy employment behaviors one year after program enrollment?
  Items measured include:
  1 item: yes (1) or no (0) questions for having a resume (dichotomous) Yes responses indicate employment readiness, so the higher the rating, the better the score.
Time Frame: Change from baseline in father financial behavior at 12 months from enrollment.]
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Services
Number analyzed (Participants) | 158
Participants
  have resume at baseline | 24
  have resume at follow-up | 97

7. Secondary Outcome: Healthy Employment Attitudes
Description: Will Fresno Fatherhood program participants experience significant increases in healthy employment attitudes/beliefs/expectations after completing the Fresno Fatherhood program?
  Items measured include:
  8 items: levels of agreement with key employment attitudes (categories, 5-point scale)
  1. Strongly Disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly Agree
  The 8 items are measured as a construct. All items are added together and divided by 8 to create the construct score. The higher the score, the better the outcome.
  maximum score of 5.0, minimum score of 1.0
Time Frame: Change from baseline in healthy employment attitudes to immediately after program completion.
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | Primary Services
Number analyzed (Participants) | 413
score on scale
  mean at baseline | 3.97 (.660)
  mean at follow-up | 4.09 (.620)

ADVERSE EVENTS:
Time Frame: 1 year through study completion
Description: The definitions of adverse events do not differ from the clinicaltrials.gov definitions.
Arm/Group | Primary Services
All-Cause Mortality (participants affected / at risk) | 0/488
Serious Adverse Events (participants affected / at risk) | 0/488
Other Adverse Events (participants affected / at risk) | 0/488

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT05239754/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-16): https://cdn.clinicaltrials.gov/large-docs/54/NCT05239754/SAP_001.pdf